CLINICAL TRIAL: NCT02318901
Title: A Phase Ib/II Study of Pembrolizumab and Monoclonal Antibody Therapy in Patients With Advanced Cancer (PembroMab
Brief Title: Pembrolizumab and Monoclonal Antibody Therapy in Advanced Cancer
Acronym: PembroMab
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI no longer at sight. Results not collected
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PembroMab
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Advanced Cancer; Breast Cancer; Gastric Cancer; Esophageal Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms | interventions — pembrolizumab; Trastuzumab; Ado-Trastuzumab Emtansine; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. Intravenous (i.v.) trastuzumab 6 mg/kg on day 1 every 21 days.
  Interventions: Drug: Pembrolizumab; Drug: Trastuzumab
- Arm 2 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. i.v. ado-trastuzumab emtansine 3.6 mg/kg on day 1 every 21 days.
  Interventions: Drug: Pembrolizumab; Drug: ado-trastuzumab emtansine
- Arm 3 (Experimental): Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. i.v. cetuximab 400 mg/m2 on cycle 1 day 1, then i.v. cetuximab 250 mg/m2 on day 8. Each subsequent cycle will be i.v. cetuximab 250 mg/m2 on days 1 and 8 every 21 days.
  Interventions: Drug: Pembrolizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: KEYTRUDA
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Arm 1
Drug: ado-trastuzumab emtansine
  Other Names: Kadcyla
  Arms: Arm 2
Drug: Cetuximab
  Other Names: Erbitux
  Arms: Arm 3

SUMMARY:
There will be two phase II cohorts for pembro plus trastuzumab: one cohort will be for patients with unresectable HER2 overexpressing gastric or GEJ cancers, the other cohort will be for patients with HER2 overexpressing metastatic breast cancer (MBC). The pembro plus ado-trastuzumab emtansine phase II arm will be for patients with HER2 overexpressing MBC. There will be two phase II cohorts for pembro plus cetuximab: one cohort will be for patients with HNSCC, the other cohort will be for patients with K-ras, B-raf, N-ras wildtype metastatic CRC.

DETAILED DESCRIPTION:
Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. Pembrolizumab will be infused prior to the start of the assigned monoclonal antibody (Mab) arm. .

Dosing for the Mab arms will begin as follows:

Arm 1: Cycle length is 21 days. Intravenous (i.v.) trastuzumab 6 mg/kg on day 1 every 21 days.

Arm 2: Cycle length is 21 days. i.v. ado-trastuzumab emtansine 3.6 mg/kg on day 1 every 21 days.

Arm 3: Cycle length is 21 days. i.v. cetuximab 400 mg/m2 on cycle 1 day 1, then i.v. cetuximab 250 mg/m2 on day 8. Each subsequent cycle will be i.v. cetuximab 250 mg/m2 on days 1 and 8 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has definitive histologically or cytologically confirmed unresectable or metastatic solid tumor.
2. Patient has one or more tumor measurable as defined by RECIST 1.1 by CT scan (or PET/CT, if patient is allergic to CT contrast media).
3. Patients can be enrolled only on one of the treatment arms on this trial.
4. The investigator will select the appropriate treatment arm for the patient with the following requirements: (a) Patients cannot have had prior progression or intolerance to a specific Mab and then enrolled on an arm with that same Mab plus pembro, (b) The Mab on the arm selected must be considered standard of care or listed in the NCCN guidelines (www.nccn.org) for that cancer type. For Arm 1, patients with HER2 overexpressing MBC eligible for maintenance trastuzumab are allowed after taxane plus trastuzumab plus pertuzumab combination therapy.
5. Have recovered from acute toxicities of prior treatment:

   1. > 3 weeks must have elapsed since receiving any investigational agent.
   2. > 2 weeks must have elapsed since receiving any radiotherapy, or ≥ 3 weeks or 5 half-lives whichever is shorter for treatment with cytotoxic or biologic agents ( ≥ 6 weeks for mitomycin or nitrosoureas). Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted.
6. Patient has adequate biological parameters as demonstrated by the following blood counts at time of screening:
7. Absolute neutrophil count (ANC) > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 9 g/dL.
8. Serum creatinine ≤2.0, total bilirubin ≤ 2 mg/dL, AST/ALT ≤ 5 times the upper limit of normal (ULN) range
9. Thyroid stimulating hormone (TSH) within institutional normal limits. If TSH is above the upper limit of normal range, then a free T4 within institutional normal limits is acceptable.
10. Persistent prior systemic therapy non-hematologic AE grade ≥ 2 (except alopecia or correctable electrolyte abnormality with supplementation)
11. Patient has a Karnofsky performance status (KPS) ≥ 70.
12. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial.

Inclusion criteria for Phase II only:

1. Patients must have unresectable HER2 overexpressing gastric or GEJ cancers to be enrolled on Cohort 1 of the pembro plus trastuzumab phase II portion.
2. Patients must have HER2 overexpressing MBC to be enrolled on Cohort 2 of the pembro plus trastuzumab phase II portion.
3. Patients must have HER2 overexpressing MBC to be enrolled on pembro plus ado-trastuzumab emtansine phase II portion.
4. Patients must have HNSCC to be enrolled on Cohort 1 of the pembro plus cetuximab phase II portion.
5. Patients must have K-ras, B-raf, N-ras wildtype CRC to be enrolled on Cohort 2 of the pembro plus cetuximab phase II portion.

Exclusion Criteria:

1. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
2. Serious non-healing wound, ulcer, or bone fracture.
3. Patient has known brain metastases, unless previously treated and well-controlled for at least 1 month (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
4. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
5. Patient has known active infection with HIV, hepatitis B, or hepatitis C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol).
6. Requiring daily corticosteroid dose ≥ 10 mg prednisone or equivalent per day.
7. Patient has undergone major surgery, other than diagnostic surgery (e.g., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
8. Patient has a history of allergy or hypersensitivity to any of the study drugs or any of their excipients, or the patient exhibits any of the events outlined in the Contraindication or Special Warnings and Precautions sections of the product or comparator SmPC or Prescribing Information.
9. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
10. Patient will be receiving any other anti-cancer therapy during participation in this trial.
11. Prior treatment with pembro. Receipt of other PD-1 inhibitors or PD-L1 inhibitors is allowed.
12. Active or prior documented autoimmune disease requiring systemic treatment within the past 2 years.

Exclusion Criteria for phase II portion only:

1. Patients with a history of more than one primary cancer, with the exception of: a) curatively resected nonmelanomatous skin cancer; b) curatively treated cervical carcinoma in-situ; or c) other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the 2 years prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, FNP, Study Director — Western Regional Medical Center; Alan Tan, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center/Cancer Treatment Center of America, Goodyear, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. Intravenous (i.v.) trastuzumab 6 mg/kg on day 1 every 21 days.
  Pembrolizumab
  Trastuzumab
- Arm 2: Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. i.v. ado-trastuzumab emtansine 3.6 mg/kg on day 1 every 21 days.
  Pembrolizumab
  ado-trastuzumab emtansine
- Arm 3: Pembrolizumab 2mg/kg administered intravenously over 30 minutes every 3 weeks. i.v. cetuximab 400 mg/m2 on cycle 1 day 1, then i.v. cetuximab 250 mg/m2 on day 8. Each subsequent cycle will be i.v. cetuximab 250 mg/m2 on days 1 and 8 every 21 days.
  Pembrolizumab
  Cetuximab
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 5 | 1 | 10
Completed | 0 | 0 | 0
Not Completed | 5 | 1 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 5 | 1 | 10 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 10 | 16
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 52 [44 to 64] | 62 | 58 [35 to 67] | 57 [35 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 10 | 11
  Male | 4 | 1 | 0 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 1 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Determine the Recommended Phase 2 Dose (RP2D) of Monoclonal Antibody Therapy (Mab) in Combination With Pembrolizumab (Pembro) in Subjects With Advanced Cancer
Description: PI left site. Study was prematurely terminated. No additional study items were conducted including, data collection, results or statistical analysis completed.
Time Frame: 3 weeks
Population: PI left site. Study was prematurely terminated. No additional study items were conducted including, data collection, results or statistical analysis completed.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Frequency of Grade 3 or Higher Treatment-related Adverse Events by CTCAE 4.03
Description: as for outcome 1
Time Frame: up to 12 months
Population: No data was analyzed for this trial. PI left site unexpectedly.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Response Rate by irRC and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria
Description: as for outcome 1
Time Frame: 12 weeks
Population: No data was analyzed for this trial. PI left site unexpectedly.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: To Determine the Overall Survival (OS) and Progression-free Survival (PFS)
Description: as for outcome 1
Time Frame: up to 12 months
Population: No data was analyzed for this trial. PI left site unexpectedly.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: To Characterize Changes in Circulating Tumor DNA in Patients Enrolled on This Study
Description: as for outcome 1
Time Frame: up to 12 months
Population: No data was analyzed for this trial. PI left site unexpectedly.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Textural Changes Identified on Imaging That is Done Per Routine Practice
Description: as for outcome 1
Time Frame: 12 weeks
Population: No data was analyzed for this trial. PI left site unexpectedly.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: PI no longer at site. Results not collected
Description: PI no longer at site. Results not collected
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT02318901/Prot_SAP_000.pdf